CLINICAL TRIAL: NCT05977348
Title: Increasing Food Literacy as a Means of Increasing Preschool Children's Food Acceptance and Reducing Obesity Risk
Brief Title: Increasing Food Literacy in Preschoolers to Reduce Obesity Risk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Lori Francis, Professor of Biobehavioral Health, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OSP#233045; 2023-68015-39416 (Other Grant/Funding Number: United States Department of Agriculture)
Record Dates: First submitted 2023-07-18; First posted 2023-08-04 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Food Preferences; Food Selection; Eating, Healthy; Obesity, Childhood
Keywords: Food literacy; Healthy growth; Child Development; Food Acceptance
MeSH Terms: conditions — Food Preferences; Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: The project is a cluster-randomized trial, with a 1:1 ratio of classroom random assignment to intervention or control.
Who Masked: Outcomes Assessor
Masking Description: Study team members who will conduct individual research assessments with each child will be blinded to study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Bodies Project Comparison (HBP) (No Intervention): All classrooms will receive the Eating the Alphabet curriculum, which includes 27 lessons that introduce children to a new fruit or vegetable from A-Z each week. Parents in comparison and intervention classrooms will receive access to web-based parent resources related to the Eating the Alphabet curriculum (e.g., food of the week fact sheets with recipes and suggestions for use, and coloring pages).
- Healthy Bodies Project Plus (HBP+) (Experimental): Intervention classrooms will receive the Eating the Alphabet curriculum described above for comparison classrooms, in addition to (1) the Healthy Eating curriculum, (2) classroom materials and teacher training designed to improve the classroom food and mealtime environment in ways that increase food acceptance, and (3) parent/caregiver education on responsive food parenting.
  Interventions: Behavioral: Healthy Eating Curriculum; Behavioral: Improving the Classroom Food and Mealtime Environment; Behavioral: Parent Education; Behavioral: ECE Food Acceptance Training

INTERVENTIONS:
Behavioral: Healthy Eating Curriculum — The Healthy Eating (HE) curriculum is designed to provide children with skills needed to develop healthy eating habits. Each lesson builds upon the overall goal of creating a healthy restaurant. Children are taught to identify differences between GO and WHOA foods, recognize the five food groups, and learn to make healthy food choices.
  Arms: Healthy Bodies Project Plus (HBP+)
Behavioral: Improving the Classroom Food and Mealtime Environment — HBP+ Classrooms will receive additional sensory activities for each lesson (e.g., posters, food models, games) designed to improve the classroom food environment and provide repeated exposure to activities and messages about fruits and vegetables. Teachers in HBP+ classrooms will be provided with additional training on strategies shown to increase food acceptance in preschool children (e.g., modeling, encouraging children to try foods without coercion). In addition, HBP+ classrooms will include "tasting charts" that children will stamp to indicate their liking for each food each week.
  Arms: Healthy Bodies Project Plus (HBP+)
Behavioral: Parent Education — Parents in intervention classrooms will be given access to 8 web-based lessons on food parenting and responsive parenting. Topics include: establishing mealtime routines, shopping healthy on a budget; modeling of healthy eating behaviors; addressing picky eating in children; structuring low-stress mealtime environments; the division of responsibility in feeding, and portion control.
  Arms: Healthy Bodies Project Plus (HBP+)
Behavioral: ECE Food Acceptance Training — HBP+ early childhood educators (ECEs) will be asked to complete an online, self-paced course on increasing food acceptance in preschool children. Topics will include: repeated exposure to foods; modeling of healthy eating behaviors; addressing picky eating in children; structuring low-stress mealtime environments; and the division of responsibility in feeding.
  Arms: Healthy Bodies Project Plus (HBP+)

SUMMARY:
The goal of this clinical trial is to examine the effects of a nutrition education program on preschool children's food literacy and food acceptance, and to examine the added influence of a healthy eating curriculum and parent education on children's food knowledge and healthful food choices. The project will be evaluated with 450 children ages 3 to 5 years in center-based childcare programs serving predominantly Supplemental Nutrition Assistance Program (SNAP)-eligible families in Pennsylvania. Outcomes for children who receive the added healthy eating curriculum will be compared to children in classrooms that only receive the nutrition education program.

DETAILED DESCRIPTION:
Repeatedly exposing young children to new foods can increase their willingness to try those foods, and they may - with time - learn to like those foods. Being able to learn about, touch and taste new foods can be a powerful tool to foster young children's liking of new foods. This project's goals are to test whether a preschool nutrition education program can improve (1) children's ability to name and identify fruits and vegetables, (2) children's knowledge about food and nutrition, (3) children's healthful food choices during a meal, and (4) parenting around children's eating. Participants will include 450 children ages 3 to 5 years in center-based childcare programs serving a large majority of families experiencing poverty in Pennsylvania. In all classrooms, children will receive food literacy lessons designed to help them learn about different fruits and vegetables, where they grow, and why they are good for our bodies. Children in intervention classrooms will receive food literacy lessons, in addition to lessons on healthy eating designed to improve children's nutrition knowledge. Teachers in intervention classrooms will be provided with materials designed to increase children's knowledge about nutrition and healthy eating. Intervention parents will receive web-based lessons designed to improve parenting practices related to children's eating behaviors. The study will be conducted over a 14-month period, and a variety of child, teacher, classroom and parent outcomes will be measured before, during and after the intervention. The results of this study are anticipated to add new information on ways to improve children's nutrition knowledge and acceptance of fruits and vegetables.

ELIGIBILITY:
Inclusion Criteria:

* Preschool children enrolled in participating centers

Exclusion Criteria:

* Severe food allergies that prevent children from consuming project foods
* Presence of a developmental or sensory disability that affects food intake and/or learning
* Lack of English fluency (children and caregivers)
* Children not regularly present during days/times that intervention lessons are delivered
* Parents who are not involved in feeding/preparing meals for children at least 50% of the time

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 770 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Children's Food Acceptance | Change from baseline to post-intervention (~6 months)
  Teachers reports of each child's willingness to try and liking of weekly target foods; lab-created measure. Scores for trying (yes/no) and liking (yes/no) are summed to create total scores for each. Scores range from 0 to 26 for trying and liking. Higher scores indicate a higher frequency of trying weekly foods and higher frequency of liking seeking foods.
Children's willingness to try novel foods | Change from baseline to post-intervention (~6 months)
  Observed measure of children's willingness to try 4 novel foods (The Tasting Game; lab-created measure). The child scores 1 point for each bite of food that is tasted or eaten. Scores for each range from 0 (none tasted/eaten) to 3 (all pieces tasted/eaten). Total scores range from 0 to 12, and are created by summing the points obtained for each food item. Higher scores indicate a greater willingness to try foods.
Children's Food Literacy | Change from baseline to post-intervention (~6 months)
  Observed measure of children's ability to name/identify 6 foods using pictures (Food Literacy Scale; lab-created measure). Children receive a score of 0 (incorrect/don't know), 1 (correctly identified on the second pass), or 2 (correctly named on the first pass) points. Total scores range from 0 to 12, and are created by summing the points obtained for each food item. Higher scores indicate higher food literacy or ability to identify foods.
Children's Food Knowledge | Change from baseline to post-intervention (~6 months)
  Observed measure of children's ability to differentiate between nutrient- and energy-dense foods using the Snack Selection Protocol (Sigma-Grant et al., 2014). Children receive 1 point for each nutrient-dense food item chosen. Scores range from 0-18, with higher scores indicating nutrient-dense foods being chosen more often energy-dense foods.
Children's Food Choices | Change from baseline to post-intervention (~6 months)
  Observed measure of children's food choices when given the option to choose a nutrient- vs. energy-dense snack (live-coded; lab-created measure). Children receive a score of either 0 (energy-dense food chosen) or 1 (nutrient-dense food chosen).

SECONDARY OUTCOMES:
Child Weight Status/Adiposity | Change from baseline to post-intervention (~6 months)
  Child age- and sex-specific Body Mass Indices (BMI) from measured height and weight. Conditional weight gain (rate of change in children's BMIz), will be calculated as the standardized residual of the linear regression of post-intervention BMIz predicted by baseline BMIz, adjusted for child age and sex.

OTHER OUTCOMES:
Child food requests (parent report) | Change from baseline to post-intervention (~6 months)
  Children's requests for foods used in the study, as well as general requests for fruits and vegetables (Fruit and Vegetable Survey; lab-created measure).
Children's Appetitive Traits and Behaviors (parent and teacher report) | Baseline
  Measure of food approach and avoidance behaviors (e.g., satiety responsiveness and food enjoyment) measured using the Children's Eating Behaviour Questionnaire (Wardle et al., 2001). Response options range from 1 to 5 and subscale scores are calculated by averaging the items within each subscale. Higher scores for any subscale indicate the respondent's perception of a greater degree of the particular eating style in the child.
Children's Food Exposure (parent and teacher report) | Baseline
  Measure of children's previous experience and familiarity with target foods using the Children's Food Exposure Questionnaire (lab-created). Scores are calculated by averaging the items within each subscale. Subscale 1 scores range from 0-8 points, subscales 2-6 scores range from 0-3. Higher scores for subscales indicate (1) higher availability of fruits and vegetables; (2) more encouragement to eat fruits and vegetables; (3) more modeling of fruit and vegetable consumption by mothers; (4) more asking for fruits and vegetables by children; (4) children have more barriers to eat fruits and vegetables; (6) and caregivers have more barriers to eat fruits and vegetables respectively.
Children's Mealtime Behaviors | Change from baseline to post-intervention (~6 months)
  A lab-created, parent-report measure of children's media use while eating. Response options on this 3-item measure range from 1 to 4. Scores are calculated by averaging the items, with higher scores indicate a higher frequency of the child eating while watching television.
Food parenting practices (parent-report) | Change from baseline to post-intervention (~6 months)
  Measure of parents' food-related practices (e.g., coercive vs. responsive feeding practices) using the Comprehensive Feeding Practices Questionnaire (Musher-Eizenman & Holub, 2007). This instrument includes 12 sub scales with response options ranging from 1-5; items are averaged to create each sub scale. Higher scores indicate a greater degree or frequency of use of the food parenting strategy.
Parent Nutrition Knowledge | Change from baseline to post-intervention (~6 months)
  Parent/caregiver knowledge about topics such as appropriate portion sizes, number of snacks preschoolers need each day, etc. using an adapted version of a Nutrition Knowledge Questionnaire developed by Rapson et al. (2020). This adapted 53-item questionnaire includes forced-choice and open-ended questions. Respondents score 1 point for correct answers on all nutrition knowledge items and 0 points for an incorrect or "choose not to answer" response. Incorrect responses, or responses that are contradictory to nutrition guidelines are also scored as 0 points. A composite score is obtained by summing answers to all nutrition knowledge items. Higher scores indicate a higher levels of nutrition knowledge to support healthy eating/feeding practices for preschool aged children.
Household Food Security (parent-report) | Baseline
  Household, adult and child food insecurity and hunger measured using the 18-item U.S. Household Food Security Survey. If there is no missing data, respondents can be categorized based on their sum score across all 18 questions. Categories and their respective scores are as follows: (1) High Food Security: 0-2 points, (2) Marginal Food Security: 3-7 points, (3) Low Food Security: 8-12 points, and (4) Very Low Food Security: 13-18 points. Affirmative items (with responses) are summed to create a raw score, with scores ranging from 0-18 points. Higher scores indicate greater household food insecurity.
Household Demographics and Parents' General Health (parent-report) | Baseline
  Sociodemographic information, parent height and weight (lab-created questionnaire).
Childcare Provider Nutrition Knowledge | Change from baseline to post-intervention (~6 months)
  Childcare provider knowledge about topics such as appropriate portion sizes, number of snacks preschoolers need each day, etc. measured using an Early Childhood Educator Nutrition Knowledge Questionnaire developed by Rapson et al. (2020). This 57-item questionnaire includes forced-choice and open-ended questions. Respondents score 1 point for correct answers on all nutrition knowledge items and 0 points for an incorrect or "choose not to answer" response. Incorrect responses, or responses that are contradictory to nutrition guidelines are also scored as 0 points. A composite score is obtained by summing answers to all nutrition knowledge items. Higher scores indicate a higher levels of nutrition knowledge to support healthy eating/feeding practices for preschool aged children.
Childcare Provider Feeding Beliefs | Change from baseline to post-intervention (~6 months)
  Childcare provider mealtime behaviors and feeding practices measured using the About Feeding Children questionnaire (Swindle et al., 2018). This questionnaire contains 31 items and 9 subscales. Higher scores on each of the subscales indicate the degree to which the respondent utilizes the mealtime strategy or agrees with particular mealtime beliefs.
Childcare Provider Demographics | Baseline
  Sociodemographic information, teaching experience, height, weight, physical activity frequency (lab-created questionnaire).
Classroom Food and Mealtime Environment | Change from baseline to post-intervention (~6 months)
  An observational measure of the classroom food and mealtime environment. Response options range from 1 to 4, and scores are calculated by averaging the items within each subscale. Higher scores indicate (1) a higher degree of visuals that support healthy eating; and (2) teacher and child dynamics during mealtime that are consistent with healthy eating practices.
Classroom Chaos | Baseline
  An adapted measure of classroom chaos using the Confusion, Hubbub and Order Scale for classrooms (Wachs et al., 2004). Response options range from 1 to 4, and a total score is calculated by averaging scores for 12 items. Higher scores indicate more chaos, disorganization, and noise level in the classroom.

CONTACTS AND LOCATIONS:
Overall Officials: Lori A Francis, Ph.D., Principal Investigator — Penn State University; Professor
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after all primary and secondary analyses are completed to address study aims.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be made available in perpetuity after all primary and secondary analyses are completed to address study aims.
Access Criteria: The data can be accessed by contacting the principal investigator after the specified time period.